CLINICAL TRIAL: NCT00939965
Title: Pilot Study to Investigate the Feasibility of 13-cis-retinoic Acid Pharmacokinetic Monitoring in High-risk Neuroblastoma Patients
Brief Title: Isotretinoin in Treating Young Patients With High-Risk Neuroblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-PK-2008-03; CDR0000637053 (Registry Identifier: PDQ (Physician Data Query)); EU-20914; EUDRACT-2008-003606-33
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Neuroblastoma
Keywords: localized unresectable neuroblastoma; recurrent neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin; Polymerase Chain Reaction

INTERVENTIONS:
Drug: isotretinoin
Genetic: DNA analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors plan better treatment for patients receiving isotretinoin.

PURPOSE: This clinical trial is studying the side effects and best dose of isotretinoin in treating young patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the feasibility of implementing individualized dosing of isotretinoin in patients with high-risk neuroblastoma after course 1 of treatment, based on isotretinoin pharmacokinetics and toxicity.
* To minimize the large inter-patient variation in plasma concentrations of isotretinoin.
* To ensure that patients are not exposed to potentially sub-optimal plasma concentrations of isotretinoin during long-term treatment, particularly for patients who are not able to swallow isotretinoin capsules.

Secondary

* To obtain preliminary data on the potential impact of isotretinoin therapeutic monitoring on clinical response and toxicity in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral isotretinoin twice daily on days 1-14. Courses repeat every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and during courses 1-3 for pharmacokinetic studies and determination of each patient's individual therapeutic-dose level requirement. Genotyping to identify genes that metabolize enzymes is conducted via PCR.

After completion of study therapy, patients are followed up periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk neuroblastoma
* Concurrent isotretinoin as part of clinical treatment

PATIENT CHARACTERISTICS:

* Not pregnant
* Fertile patients must use effective contraception
* Has a single- or double-lumen central venous catheter in place

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-02

PRIMARY OUTCOMES:
Pharmacokinetics of isotretinoin
Toxicity according to NCI CTCAE v.3

SECONDARY OUTCOMES:
Clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Veal, Principal Investigator — University of Newcastle Upon-Tyne
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital for Children, London, England
  - University of Newcastle-Upon-Tyne Northern Institute for Cancer Research, Newcastle upon Tyne, England
  - Royal Marsden - Surrey, Sutton, England